CLINICAL TRIAL: NCT04404166
Title: Phone-based Intervention Under Nurse Guidance After Stroke 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northern California Institute of Research and Education (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bruce Ovbiagele, Chief of Staff, Northern California Institute of Research and Education
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-30016; 5R01HL152188-05 (NIH)
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Blood Pressure; Stroke; Cardiovascular Diseases
MeSH Terms: conditions — Stroke; Cardiovascular Diseases | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PINGS 2 (Experimental): Participants received a 12-month, multicomponent, nurse-led intervention in addition to usual post-stroke care. The intervention included:
  Home blood pressure monitoring at least weekly with nurse follow-up for threshold breaches.
  Mobile phone medication reminders (daily alarms set on the participant's own device).
  Weekly audio health education messages in local dialects emphasizing stroke risk factor control and medication adherence.
  Nurse navigators provided case management, coordinated clinic visits as needed, and tracked blood pressure readings and adherence.
  Interventions: Behavioral: PINGS 2
- Standard of Care (Active Comparator): Participants received standard secondary prevention after stroke according to local guidelines. This typically included periodic physician follow-up, antihypertensive therapy, antiplatelets, and statins prescribed at the clinician's discretion.
  To maintain contact frequency similar to the intervention group, participants received neutral lifestyle text messages unrelated to hypertension or stroke prevention.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: PINGS 2 — Home BP monitoring, medication reminders using phone alerts, and patient education on hypertension, cardiovascular risk reduction & stroke
  Arms: PINGS 2
Other: Standard of Care — Standard of Care (routine post-stroke management per guidelines)
  Arms: Standard of Care

SUMMARY:
The overall objective of Phone-based Intervention under Nurse Guidance after Stroke II (PINGS-2) is to deploy a hybrid study design to firstly, demonstrate the efficacy of a theoretical-model-based, mHealth technology-centered, nurse-led, multi-level integrated approach to substantially improve longer term BP control among 500 recent stroke patients encountered at 10 hospitals in Ghana. Secondly, PINGS II seeks to develop an implementation strategy for routine integration and policy adoption of mhealth for post-stroke BP control in a LMIC setting. The investigators will leverage experience gained from the NIH Global Brain Disorders funded R21 pilot study (NS094033) to test efficacy of a refined, culturally-tailored, and potentially implementable intervention aimed at addressing the premier modifiable risk for stroke & other key variables in an under-resourced system burdened by suboptimal care & outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years (stroke is commoner above this age cut-off)
* male or females (sex is a biologic variable of interest)
* recent stroke (within one month of symptom onset)- stroke may be ischemic or hemorrhagic based on brain imaging or diagnosed clinically using the locally validated version of the 8-item questionnaire for verifying stroke free status (8-QVSFS) when neuroimaging is not feasible
* uncontrolled HTN (SBP ≥ 140 mmHg at both the last clinical encounter post-stroke and the eligibility screening visit) - SBP is used as the selection variable since most African hypertensives <60 years have systolic or combination systolic/ diastolic HTN and for most patients, controlling SBP also results in DBP control
* patients or family carers should own a basic mobile phone that can receive text/audio messages.

Exclusion Criteria:

- Any condition that would limit participation in follow up assessments, such as severe cognitive impairment/dementia (MMSE ≤24).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Ghana (10):
  - Ankaase Methodist Hospital, Aboaso
  - Korle Bu Teaching Hospital, Accra
  - Agogo Presbyterian Hospital, Agogo
  - Cape Coast Teaching Hospital, Cape Coast
  - Komfo Anokye Teaching Hospital, Kumasi
  - Kumasi South Hospital, Kumasi
  - Kwadaso SDA Hospital, Kumasi
  - Kwame Nkrumah University of Science and Technology, Kumasi
  - Manhyia Government Hospital, Kumasi
  - Tafo Government Hospital, Kumasi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bockarie AS, Ayisi-Boateng NK, Nguah SB, Appiah LT, Fiattor T, Afriyie-Ansah S, MacCready E, Sam VA, Mensah NA, Tagge R, Agyenim-Boateng KG, Ampofo M, Laryea R, Gyamfi RA, Amuasi JH, Arthur AA, Duah C, Opare-Addo PA, Ovbiagele B, Sarfo FS, Akpalu A. The Significance of the WHO/ISH Absolute Cardiovascular Risk Prediction Scores among Recent Stroke Survivors in Ghana-Insights from the PINGS2 multicenter study. Res Sq [Preprint]. 2025 Mar 12:rs.3.rs-6175913. doi: 10.21203/rs.3.rs-6175913/v1. PMID 40162227

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period:
  First participant enrolled: October 23, 2020 Last participant enrolled: April 21, 2023 Last participant completed follow-up: April 5, 2024
  Recruitment Locations:
  10 hospitals in Ghana (3 tertiary, 2 district, 5 primary level). Urban, peri-urban, and rural populations.
  Recruitment Setting:
  Participants identified during acute stroke hospitalization or follow-up clinics. Stroke confirmed by CT (when feasible) or validated stroke-free questionnaire (QVSFS).
Pre-assignment Details: Screened: 905 potential participants.
  Excluded (n=405):
  Did not meet eligibility criteria: 243 Declined to participate: 162
  Randomized: 500 participants
Groups:
- PINGS 2: Participants received a multicomponent, 12-month nurse-led intervention in addition to usual post-stroke care.
  Components included:
  * Home blood pressure monitoring at least once weekly with nurse navigation for threshold breaches (using Omron 10 automated monitor).
  * Mobile phone medication reminders (daily alarms set on participant's own phone).
  * Weekly health education audio messages in local dialects (1-2 minutes, delivered via telephone).
  * Nurse navigators were trained to provide case management, follow algorithms for BP thresholds, and coordinate clinic visits when needed.
- Standard of Care: Participants received standard secondary prevention after stroke, according to local guidelines.
  This typically included:
  * Physician follow-up visits approximately every 2 months.
  * Prescriptions for antihypertensive agents, antiplatelets, and statins at the clinician's discretion.
  * To balance attention, participants in this group also received generic lifestyle SMS messages not related to medication adherence, hypertension, or stroke.
Period: Overall Study
Arm/Group | PINGS 2 | Standard of Care
Started | 244 | 256
Completed | 200 | 210
Not Completed | 44 | 46

BASELINE CHARACTERISTICS:
Population: Baseline characteristics include all randomized participants who started the trial and completed baseline assessments (PINGS 2: n=244; Standard of Care: n=256; total n=500). These correspond to the 244 and 256 participants listed as 'Started' in the Participant Flow module. Twelve-month outcomes were analyzed in the subset who completed follow-up (PINGS 2: n=200; SOC: n=210), as shown in the Participant Flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | PINGS 2 | Standard of Care | Total
Number analyzed (Participants) | 244 | 256 | 500
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58 (11) | 59 (11) | 58 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 116 | 219
  Male | 141 | 140 | 281
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Ghana | 244 | 256 | 500
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 157 (18) | 158 (20) | 158 (19)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 94 (13) | 96 (15) | 95 (14)
Hemoglobin A1C [Median (Inter-Quartile Range); unit: Percent] | 6 [5 to 7] | 6 [5 to 7] | 6 [5 to 7]
NIHSS Stroke Severity [Median (Inter-Quartile Range); unit: score on a scale] — National Institutes of Health Stroke Scale (NIHSS), a standardized neurological impairment scale assessing level of consciousness, visual fields, motor strength, sensory function, language, and neglect. Scores range from 0 to 42, with higher values indicating more severe neurological deficit
  score on a scale | 3 [0 to 7] | 3 [0 to 8] | 3 [0 to 8]
Modified Rankin Scale [Median (Inter-Quartile Range); unit: score on a scale] — Modified Rankin Scale (mRS), a global functional disability scale assessing residual post-stroke functional limitations. Scores range from 0 (no symptoms) to 6 (death). Higher scores reflect worse functional status.
  score on a scale | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
Hill-Bone Adherence Score [Median (Inter-Quartile Range); unit: score on a scale] — Hill-Bone Compliance to High Blood Pressure Therapy Scale, a validated 14-item adherence scale assessing medication-taking, appointment keeping, and dietary behavior. Total scores range from 14 to 56, with higher values indicating poorer adherence (i.e., worse compliance). Total score is calculated by summing item responses.
  score on a scale | 52 [50 to 53] | 52 [50 to 53] | 52 [50 to 53]
Health Literacy Score [Median (Inter-Quartile Range); unit: score on a scale] — Health Literacy Questionnaire, a validated 9-item instrument assessing understanding of hypertension and stroke. Items 1-5 use a 4-point Likert scale and items 6-9 use a 5-point difficulty scale. Total score ranges from 0 to 15, with higher scores indicating better health literacy. Total score is computed by summing all items.
  score on a scale | 9 [7 to 10] | 8 [5 to 10] | 8 [6 to 10]
Quality of Life EQ-5D [Median (Inter-Quartile Range); unit: score on a scale] — EuroQol 5-Dimension Visual Analog Scale (EQ-5D VAS), a self-reported measure of perceived overall health status. Scores range from 0 (worst imaginable health) to 100 (best imaginable health), with higher scores reflecting better health-related quality of life.
  score on a scale | 70 [50 to 83] | 70 [50 to 80] | 70 [50 to 80]
Stroke Type [Count of Participants; unit: Participants]
  Ischemic | 168 | 164 | 332
  ICH | 45 | 58 | 103
  Hemorrhagic Transformation | 8 | 2 | 10
  Untyped | 23 | 32 | 55
Diabetes Mellitus [Count of Participants; unit: Participants] | 98 | 71 | 169
Hyperlipidemia [Count of Participants; unit: Participants] | 82 | 78 | 160
Cigarette Smoking [Count of Participants; unit: Participants] | 22 | 23 | 45
Overweight/Obesity [Count of Participants; unit: Participants] | 128 | 129 | 257
Alcohol Use (Current) [Count of Participants; unit: Participants] | 28 | 24 | 52
Antihypertensive Medications at Baseline [Count of Participants; unit: Participants] — Note that subjects may be on more than one antihypertensive medication
  Participants
    ACE Inhibitors | 51 | 65 | 116
    ARBs | 115 | 115 | 230
    Betablockers | 34 | 29 | 63
    Calcium Channel Blockers | 200 | 198 | 398
    Diuretics | 56 | 48 | 104
    Methyldopa | 21 | 19 | 40
    Alpha Blockers | 7 | 7 | 14
    Antiplatelets | 148 | 151 | 299
    Statins | 176 | 186 | 362

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Target goal of <140/90 mmHg measured at baseline, months 3, 6, 9 and 12. Measured by blinded evaluator using an automated BP monitor.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Standard of Care: Usual post-stroke care per Ghanaian guidelines, including physician visits and prescriptions for secondary prevention. Received neutral lifestyle text messages unrelated to hypertension or stroke.
Arm/Group | PINGS 2 | Standard of Care
Number analyzed (Participants) | 200 | 210
participants | 67 [61 to 73] | 43 [37 to 49]
Statistical Analysis 1: Comparison: PINGS 2 vs Standard of Care; Null hypothesis: no difference in the proportion achieving SBP <140 mmHg at 12 months between PINGS 2 and Standard of Care. Analysis conducted using an intention-to-treat approach. Clinic blood pressure was measured by blinded assessors using an automated validated device. Two-sided α=0.05 was used for hypothesis testing. This outcome was prespecified as the single primary endpoint; no multiplicity adjustment was applied; Test type: Superiority — Comparison of proportions between groups using a chi-square test; two-sided α=0.05; p < 0.001, Chi-squared — Comparison of proportions (PINGS 2 vs Standard of Care), ITT population; Two-sided α=0.05; single primary endpoint, no multiplicity adjustment; Risk Difference (RD) = 24, 95% CI 2-sided [15 to 33] — The estimation parameter is the risk difference (PINGS minus Standard of Care) with corresponding 95% confidence interval

2. Secondary Outcome: Self-management
Description: Hypertension Self-Care Profile (HBP-SCP) Total Score, a validated measure assessing hypertension self-management across three domains: behavior, motivation, and self-efficacy. Each subscale ranges from 20 to 80, yielding a total score range of 60 to 240. Higher scores indicate better self-care. Month 12 total scores are reported.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale (60-240)
Arm/Group | PINGS 2 | Standard of Care
Number analyzed (Participants) | 200 | 210
score on a scale (60-240) | 100 (22) | 103 (24)
Statistical Analysis 1: Comparison: PINGS 2 vs Standard of Care; The null hypothesis was that mean self-management scores (HBP SCP) would not differ between the PINGS 2 intervention and Standard of Care at 12 months. Power calculations were based on detecting a clinically meaningful difference in systolic blood pressure, the primary outcome; this secondary outcome was exploratory; Test type: Superiority; p = 0.14, t-test, 2 sided — Unadjusted analysis comparing mean HBP SCP scores at 12 months between PINGS 2 and Standard of Care. Adjustment for baseline imbalances (stroke type and diabetes status) did not materially change the result; Mean Difference (Net) = -3.5, 95% CI 2-sided [-8.3 to 1.2] — Negative value indicates lower mean self-management score in PINGS 2 vs Standard of Care

3. Secondary Outcome: Number of Cardiovascular ED Encounters and Re-hospitalizations
Description: To be assessed via once monthly calls to patients and/or carers over 12 months of follow up in both the PINGS and usual care groups.
  Patient carers in both arms will also be encouraged to contact study team within 48 hours of hospitalizations for prompt and blinded adjudication of all potential CVD ED encounters to minimize reporting bias between the two groups.
Time Frame: 12 months
Population: All PINGS 2 completers were analyzed.
Measure: Number; unit: participants
Arm/Group | PINGS 2 | Standard of Care
Number analyzed (Participants) | 200 | 210
participants | 1 | 2
Statistical Analysis 1: Comparison: PINGS 2 vs Standard of Care; Null: no difference between arms in participants with ≥1 cardiovascular ED encounter or re-hospitalization over 12 months. Per-protocol analysis; Test type: Superiority; p = 0.9, Fisher Exact; Two-sided α=0.05; Risk Difference (RD) = -0.5 — RD = PINGS - SOC (1/200 vs 2/210)

4. Secondary Outcome: Number of Major Adverse Cardiovascular Events
Description: Major Adverse Cardiovascular events (MACE) to be assessed include recurrent stroke: fatal/ severely disabling stroke or non-fatal stroke; Coronary Artery Disease: Acute STEMI/NSTEMI, sudden cardiac deaths. MACE will be confirmed by a blinded adjudicator by reviewing where available clinical notes supported by investigations e.g. CT scan, EKGs, review of death certificates or verbal autopsy if death occurs outside hospital.
Time Frame: 12 months
Population: All PINGS 2 participants were analyzed (both completers and non completers)
Measure: Number; unit: participants
Arm/Group | PINGS 2 | Standard of Care
Number analyzed (Participants) | 244 | 256
participants | 16 | 12
Statistical Analysis 1: Comparison: PINGS 2 vs Standard of Care; Null: no difference in proportion of participants experiencing ≥1 MACE during 12-month follow-up. Events adjudicated blindly; Test type: Superiority; p = 0.5, Chi-squared; Two-sided α=0.05. No adjustment for multiple comparisons; Risk Difference (RD) = 1.9, 95% CI 2-sided [-2.6 to 6.3] — Risk difference = PINGS - SOC (16/244 vs 12/256)

5. Secondary Outcome: Health-related Quality of Life: The Euro Quality of Life-5D Questionnaire
Description: The EQ-5D questionnaire,186 will assess state of health of study participants at baseline and Month 12. Scores range from 0 (the worst possible health status) to 100 (the best possible health status).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Score on a scale (0-100)
Arm/Group | PINGS 2 | Standard of Care
Number analyzed (Participants) | 200 | 210
Score on a scale (0-100) | 76 (24) | 76 (24)
Statistical Analysis 1: Comparison: PINGS 2 vs Standard of Care; Null: no difference in mean EQ-5D scores between arms at 12 months. Secondary/exploratory outcome; power based on primary endpoint; Test type: Superiority; p = 0.9, t-test, 2 sided; Unadjusted comparison of mean EQ-5D scores (α=0.05); Mean Difference (Net) = 0.3, 95% CI 2-sided [-4.4 to 5], Standard Deviation 24 — Mean difference = PINGS - SOC; higher scores represent better quality of life

6. Secondary Outcome: Medication Adherence: Hill-Bone Compliance Scale
Description: Hill-Bone Compliance to High Blood Pressure Therapy Scale, a validated 14-item measure assessing adherence to antihypertensive therapy across three domains: medication-taking behavior, appointment keeping, and salt intake. Total scores range from 14 to 56, with higher scores indicating worse adherence (greater non-adherence). Month 12 total scores are reported.
Time Frame: 12 months
Population: participants with Month 12 data / completed follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale (14-56)
Arm/Group | PINGS 2 | Standard of Care
Number analyzed (Participants) | 200 | 210
score on a scale (14-56) | 51.5 (2.9) | 51.2 (3.7)
Statistical Analysis 1: Comparison: PINGS 2 vs Standard of Care; Null hypothesis: no difference in mean Hill-Bone adherence scores between PINGS 2 and Standard of Care at 12 months. Secondary, exploratory outcome; analysis conducted using the intention-to-treat population; Test type: Superiority; p = 0.4, t-test, 2 sided — Unadjusted comparison of 12-month mean Hill-Bone scores; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.34 to 0.93] — Mean difference calculated as PINGS 2 minus Standard of Care

7. Secondary Outcome: Medication Adherence: Medication Possession Ratio (MPR)
Description: Medication Possession Ratio (MPR), calculated as the percentage of days covered by filled antihypertensive prescriptions over 12 months. Values range from 0% to 100%, with higher values indicating better adherence. Month 12 MPR values are reported.
Time Frame: 12 months
Population: MPR collected for all randomized participants.
Measure: Mean (Standard Deviation); unit: percentage %
Arm/Group | PINGS 2 | Standard of Care
Number analyzed (Participants) | 244 | 256
percentage % | 83 (22) | 85 (21)
Statistical Analysis 1: Comparison: PINGS 2 vs Standard of Care; Null hypothesis: no difference in mean Medication Possession Ratio (MPR) between PINGS 2 and Standard of Care at 12 months. Secondary exploratory outcome; analysis conducted using the intention-to-treat population; Test type: Superiority — mean difference based on those with Month 12 MPR available; p = 0.4, t-test, 2 sided — Unadjusted comparison of 12-month mean MPR between arms (α=0.05); Mean Difference (Net) = -1.9, 95% CI 2-sided [-6.4 to 2.6] — Difference calculated as PINGS 2 minus Standard of Care

8. Other Pre Specified Outcome: Health Literacy in HPT/Stroke
Description: Self-Report: HTN/stroke Knowledge questionnaire (r=.70) Health literacy questionnaire (r = .74, .82) Assessed at months 0, 6,12. Higher scores indicate higher health literacy. Scales 1-5 are scored on a 4-point Likert-type response scale (strongly disagree, disagree, agree, strongly agree) and scales 6-9 are scored on a 5-point Likert-type scale with response options focusing on difficulty (cannot do or always difficult, usually difficult, sometimes difficult, usually easy, always easy). Month 12 is reported.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Score on a scale (0-15)
Arm/Group | PINGS 2 | Standard of Care
Number analyzed (Participants) | 200 | 210
Score on a scale (0-15) | 10 (2) | 9 (2)
Statistical Analysis 1: Comparison: PINGS 2 vs Standard of Care; Null hypothesis: no difference in mean health literacy scores between PINGS and SOC at 12 months; Test type: Superiority; p = 0.14, t-test, 2 sided; Unadjusted comparison, α=0.05; Mean Difference (Net) = 0.34, 95% CI 2-sided [-0.11 to 0.78], Standard Deviation 2 — Mean difference = PINGS - SOC; higher scores indicate better health literacy

9. Other Pre Specified Outcome: Disability/Functional Status
Description: Functional status after stroke will be assessed by Research Assistants using the Modified Rankin Scale with a scores ranging from 0 to 6, where 0=no functional limitation and 6 = death. Assessed at months 0, 3, 6, 9 and 12.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Score on a scale (0-6)
Arm/Group | PINGS 2 | Standard of Care
Number analyzed (Participants) | 200 | 210
Score on a scale (0-6) | 1.5 (1.3) | 1.6 (1.3)
Statistical Analysis 1: Comparison: PINGS 2 vs Standard of Care; Null: no difference in mean mRS scores between PINGS and SOC at 12 months; Test type: Superiority; p = 0.6, t-test, 2 sided; Unadjusted comparison; α=0.05; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.32 to 0.19], Standard Deviation 1.3 — Mean difference is PINGS - SOC; negative values favor PINGS (lower disability)

10. Other Pre Specified Outcome: Sex, Cultural, Socio-economic Factors, Study Site
Description: Assessed based on self reports at baseline. Cultural factors to assess include language spoken at home, religious observances, acceptance of gender roles; occupation, religious beliefs and dietary practices.
Time Frame: Baseline
Measure: Number; unit: Participants
Arm/Group | PINGS 2 | Standard of Care
Number analyzed (Participants) | 244 | 256
Participants
  Sex (Female) | 103 | 116
  Education (Primary or less) | 112 | 140
  Income (GHS less than or equal to 500) | 210 | 223
  Religion (Christianity) | 221 | 227
  Language Home (Akan) | 168 | 172
  Occupation (Informal/Self-employed) | 153 | 160
  Study site level (Tertiary) | 73 | 77
  Study stie level (Primary/Secondary) | 171 | 179

11. Other Pre Specified Outcome: Baseline Age
Description: Mean age of participants at enrollment, reported in years. Age is a continuous baseline characteristic and is therefore reported separately from categorical sociodemographic variables. Higher values indicate older age.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: years
Arm/Group | PINGS 2 | Standard of Care
Number analyzed (Participants) | 244 | 256
years | 58 (11) | 59 (11)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events were actively monitored throughout the 12-month follow-up period during scheduled visits at months 1, 3, 6, 9, and 12, and through monthly phone contact.
  Serious adverse events were defined according to ICH-GCP as events resulting in death, life-threatening condition, hospitalization, disability, or congenital anomaly.
  Non-serious events were recorded if reported by participants or caregivers.
Arm/Group | PINGS 2 | Standard of Care
All-Cause Mortality (participants affected / at risk) | 14/244 | 14/256
Serious Adverse Events (participants affected / at risk) | 27/244 | 18/256
Other Adverse Events (participants affected / at risk) | 0/244 | 0/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PINGS 2 (N=244) | Standard of Care (N=256)
Death (All-cause) (General disorders) | 14 | 14 — Includes all-cause mortality during 12-month follow-up.
Hospitalization (General disorders) | 7 | 3 — Hospital admissions unrelated to recurrent stroke, including infections, cardiovascular and metabolic complications.
Recurrent Stroke (Nervous system disorders) | 6 | 3 — Includes fatal, disabling, or non-fatal recurrent strokes confirmed by imaging or adjudication.
Sudden Cardiac Death (Cardiac disorders) | 10 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT04404166/Prot_SAP_000.pdf